CLINICAL TRIAL: NCT02334735
Title: Poly-ICLC Matured DC as an Adjuvant for NY-ESO-1 and Melan-A/MART-1 Peptide Vaccination Compared to Montanide® ISA-51 VG, in Study Subjects With Melanoma in Complete Clinical Remission But at High Risk of Disease Recurrence
Brief Title: A Comparison of Matured Dendritic Cells and Montanide® in Study Subjects With High Risk of Melanoma Recurrence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nina Bhardwaj (Other)
Collaborators: NYU Langone Health (Other); Memorial Sloan Kettering Cancer Center (Other); Ludwig Institute for Cancer Research (Other); Melanoma Research Alliance (Other); Oncovir, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Nina Bhardwaj, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 14-0780
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Melanoma
Keywords: Melanoma; Immunotherapy; DC Vaccine; Adjuvant Therapy; Immunogenicity
MeSH Terms: conditions — Melanoma | interventions — lentiviral minigene vaccine of COVID-19 coronavirus; poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DC Vaccine (Experimental): Study subjects receive KLH and NY-ESO-1 and Melan-A/MART-1 peptide-pulsed DCs:
  DCs per peptide antigen (NY-ESO-1 and Melan-A/MART-1) and KLH will be administered intracutaneous as a single vaccine product followed by a subcutaneous injection of Poly-ICLC (Hiltonol®).
  Interventions: Biological: DC Vaccine; Biological: Poly-ICLC
- Montanide Vaccine (Active Comparator): Study subjects receive KLH and NY-ESO-1 and Melan-A/MART-1 peptides and Montanide® ISA-51 VG:
  Vaccine consisting of NY-ESO-1 peptide, Melan-A/MART-1 peptide, and KLH with an oil phase containing Montanide ISA-51 VG adjuvant will be administered subcutaneously as a single vaccine product followed by a subcutaneous injection of Poly-ICLC (Hiltonol®).
  Interventions: Biological: Montanide Vaccine; Biological: Poly-ICLC

INTERVENTIONS:
Biological: DC Vaccine — DCs pulsed with 100µg/mL peptide (NY-ESO-1 and Melan-A/MART-1)
  10 to 15 x 106 DCs per peptide antigen (NY-ESO-1 and Melan-A/MART-1) (total not to exceed 50 x 10^6 cells)
  Arms: DC Vaccine
Biological: Montanide Vaccine — 250 µg peptide (NY-ESO-1 and Melan-A/MART-1) and 1.1 mL Montanide ISA-51 VG
  Arms: Montanide Vaccine
Biological: Poly-ICLC — 1.4 mg
  Other Names: Hiltonol®

SUMMARY:
Vaccine adjuvants are compounds used to increase specific immune responses to antigens, but have minimal toxicity or lasting immune effects on their own. This study investigates the use of dendritic cells as an adjuvant for NY-ESO-1 and Melan-A/MART-1 peptides compared to Montanide® in study subjects with melanoma in complete clinical remission.

DETAILED DESCRIPTION:
This is a Phase II open label, randomized two-arm study to evaluate the safety, tolerability, and immunogenicity of Poly-ICLC matured DCs as an adjuvant for NY-ESO-1 and Melan-A/MART-1 peptides (ARM A; DC Vaccine) compared to Montanide® ISA-51 VG (ARM B; Montanide Vaccine), both with systemic administration of Poly-ICLC on days 1 and 2 in study subjects with melanoma in complete clinical remission but at high-risk for disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent
* Histologic diagnosis of malignant melanoma, stages IIB-IV in radiologically confirmed complete clinical remission without clinical evidence of disease
* At least 4 weeks since surgery prior to first dosing of study agent
* Required values for initial laboratory tests:

  * Neutrophil count ≥ 1.0 x 10⁹/L
  * Platelet count ≥ 80 x 10⁹/L
  * Hemoglobin ≥ 10.0 g/dL
  * Serum creatinine ≤ 2.0 x mg/dL
  * AST/ALT ≤ 2.0 x upper limit of institutional normal
  * Serum bilirubin ≤ 2.0 x upper limit of institutional normal
* No active or chronic infection with HIV, Hepatitis B, or Hepatitis C
* ECOG performance status of ≤ 2
* Life expectancy of ≥ 6 months
* Men and women, ≥ 18 years of age
* Adequate venous access (for Leukapheresis and blood draws)

Exclusion Criteria:

* Serious illnesses, e.g., serious infections requiring antibiotics
* Previous bone marrow or stem cell transplant
* Study subjects with known chronic infection with HIV, hepatitis B or C. Testing will be performed if a study subject exhibits clinical signs of infection or to confirm a history of infection
* Study subjects with known autoimmune disease [e.g. SLE, RA] who have had significant symptoms within the past 3 years. Study subjects with vitiligo are not excluded
* Metastatic disease to the central nervous system
* Other malignancy within 3 years prior to entry into the study, except for treated early-stage melanoma or non-melanoma skin cancer, cervical carcinoma in situ, or incidental or localized prostate cancer treated with prostatectomy or radiation therapy, or stage I colon cancer. Patients with other completely resected malignancies in the prior three years and no evidence of disease will be evaluated on a case- by- case basis with eligibility determined based on discussion with the Principal Investigator.
* Prior chemotherapy or tumor vaccine therapy or biological therapy for treatment of melanoma. Subjects who received chemotherapy for the management of other malignancies are potentially eligible if the subject has not received chemotherapy in prior 5 years, remained disease free, and following discussion with and agreement by the principal investigator.
* Radiation therapy or major surgery within 4 weeks prior to first dose of study agent
* Concomitant treatment with systemic corticosteroids greater than physiologic doses. Topical (but not at the proposed vaccination sites) or inhalational steroids are permitted
* Participation in any other clinical trial involving another investigational agent within 4 weeks prior to first dose of study agent
* Pregnancy or lactation. Pregnancy is associated with considerable immune suppression and this additional parameter may interfere with the evaluation of dendritic cell induced immune responses in melanoma study subjects. Pregnancy test must be negative on all women of reproductive potential at baseline (within 7 days of entry into the study) and they must agree to use birth control measures while on the study.
* Study subjects previously treated with one of the peptides used in this trial, melanoma protein vaccine, melanoma whole cell vaccines, or with Montanide are not eligible
* Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of study agents hazardous or obscure the interpretation of AEs
* Lack of availability of study subject for immunological and clinical follow up assessments
* Children < 18 years of age
* Allergy to shellfish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Humoral immune response | up to 3 years
  Humoral immune responses will be determined by the presence of NY-ESO-1 and Melan-A/MART-1 specific antibodies by ELISA
Cytokine secretion | up to 3 years
  Cytokine secretion by NY-ESO-1 and Melan-A/MART-1 specific CD4+ and CD8+ T cells, as a measure of T cell activation, will be determined by flow cytometry analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Bhardwaj, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - New York University Langone Medical Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided